CLINICAL TRIAL: NCT05985967
Title: Therapeutic Modalities on Exercise Performance and Post-exercise Recovery of CrossFit® Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3.997.120-1
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Muscle Strength
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Control (Other): Passive recovery for 30 minutes
  Interventions: Other: Passive recovery
- PBMT-sMF (Experimental): Photobiomodulation therapy combined with static magnetic field, with a total treatment duration lasting for around 30 minutes.
  Interventions: Device: PBMT-sMF
- Shock wave (Active Comparator): Shock wave therapy applied for 30 minutes.
  Interventions: Device: Shock wave
- Pneumatic compression (Active Comparator): Pneumatic compression applied for 30 minutes.
  Interventions: Device: Pneumatic compression

INTERVENTIONS:
Device: PBMT-sMF — PBMT-sMF applied in the lower limbs with different doses per muscle group.
  Arms: PBMT-sMF
Device: Shock wave — Shock wave therapy applied in the lower limbs for 30 minutes.
  Arms: Shock wave
Device: Pneumatic compression — Pneumatic compression applied in the lower limbs for 30 minutes.
  Arms: Pneumatic compression
Other: Passive recovery — Volunteers laid in supine position resting for 30 minutes.
  Arms: Control

SUMMARY:
Crossfit® is a training modality that consists in functional movements, constantly varied and executed at high intensity. Both training sessions and competitions involve physically demanding activities, which in addition to being performed at very high intensity also involves the aerobic metabolism pathway. These characteristics led to very high metabolic and muscular stress, as well as decrease in physical performance immediately after competitions and training sessions. The cumulative effects of the metabolic and muscular stress can be a precursor of injuries. Studies using different therapeutic modalities aiming to improve post-exercise recovery are needed in order to tackle this issue.

However, to the date there are no studies investigating the effects of different therapeutic modalities in an exercise modality such as Crossfit®. Therefore, the aim of this project is to assess the effects of different therapeutic modalities on performance and muscle recovery of Crossfit® athletes.

DETAILED DESCRIPTION:
It will be carried out a randomized, crossover, controlled trial.

Volunteers will be allocated to four interventions, and the order of the interventions will be randomized.

The outcomes will be obtained at baseline (prior to the Workout of the Day - WOD), and in different timepoints after that.

The WOD will be consisted in finishing as quickly as possible a sequence of three exercises (Calories in Assault AirBike®, Hang Squat Clean and Box Jump Over), in a well-known series model for the athletes, without rest.

The investigators will analyze: the maximum number of free squats performed in 1 minute; the activity of creatine kinase (CK); the levels of Interleukin-6 (IL-6); the ratings of perceived exertion; and the volunteers satisfaction with the interventions.

All data will be analyzed both in their absolute values and in relation to their percentage variation from the values obtained in the pre-WOD (baseline) assessments.

ELIGIBILITY:
Inclusion Criteria:

* Crossfit® amateur male athletes
* Do not present a history of musculoskeletal injury in the regions of the hips, knees and calves in the month preceding the study;
* Are not using pharmacological agents;
* Athletes should have been practicing the sport for at least 1 year;
* Voluntarily commit to participate in all stages of the study.

Exclusion Criteria:

* Present musculoskeletal or joint injuries during data collection.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity | 1hour, 24 hours and 48 hours after WOD (workout of the day).
  The functional capacity will be assessed through the maximum number of free squat repetitions performed within 1 minute.

SECONDARY OUTCOMES:
Change in the activity of creatine kinase (CK) | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  The activity of CK will be analyzed from the blood samples collected from the participants through spectrophotometry and using specific reagent kits.
Change in the levels of interleukin-6 (IL-6) | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  The levels of interleukin-6 will be analyzed from the blood samples collected from the participants through enzyme-linked immunosorbent assay (ELISA) and using specific reagent kits.
Participants' perceived exercise intensity | 1 minute after WOD (workout of the day), 1 minute post-treatment/intervention, 1 hour, 24 hours and 48 hours after WOD.
  The perception of exercise intensity will be assessed through a 0-100 Ratings of Perceived Exertion Scale: in this scale lower score, means lower degree of fatigue and higher score, means higher degree of fatigue.
Participants' satisfaction regarding the interventions | 48 hours after WOD (workout of the day).
  The participants satisfaction regarding the interventions will be assessed through the LIKERT scale

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, Ph.D., Principal Investigator — Full Professor
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available six months after the manuscript publication for five years after that.
Access Criteria: All IPD that underlie results in a publication will be available on reasonable request.